CLINICAL TRIAL: NCT03923634
Title: A Prospective Open-label, Multicenter Study Evaluating Princess® RICH in Correction of Fine Lines
Brief Title: Princess® RICH for the Correction of Fine Lines
Acronym: RICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPH-401-201364
Record Dates: First submitted 2019-04-08; First posted 2019-04-22 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Lateral Canthal Lines; Perioral Rhytids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Princess® RICH (Experimental): Eligible subjects will be injected with Princess® RICH (this is an open-label study).
  Princess® RICH is injected into the lateral canthal lines and/or perioral rhytids.
  Interventions: Device: Princess® RICH

INTERVENTIONS:
Device: Princess® RICH — Princess® RICH is injected into lateral canthal lines and/or perioral rhytids

SUMMARY:
Eligible subjects deemed by the treating physician to have sufficient severity to merit treatment of either their lateral canthal lines (LCL) or perioral rhytids (PR) or both will be treated with Princess® RICH at the Baseline visit and at week 3 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Subjects deemed by the treating physician to have LCL and/or PR of sufficient baseline severity to merit treatment with Princess® RICH to be corrected
* A negative urine pregnancy test at Visit 1 and commitment to use an adequate method of birth control for the duration of the clinical investigation (for women of childbearing potential only.)
* Healthy skin in the facial area and free of diseases that could interfere in cutaneous aging evaluation
* Willingness to abstain from any aesthetic or surgical procedures in the treatment area for the duration of the clinical investigation
* Written signed and dated informed consent

Exclusion Criteria:

* Tendency to hypertrophic scars, pigment disorders or keloid formation.
* History of autoimmune disease or receiving therapy for modification of immune response
* Hypersensitivity to hyaluronic acid or glycerol.
* Permanent fillers in the areas to be treated.
* Subjects who are pregnant or breast feeding.
* Subjects who are anticoagulated or with history of bleeding disorder.
* Daily treatment with platelet aggregation inhibitors unless previously cleared by their primary care physician.
* Cutaneous, inflammatory and/or infectious processes present at V0, recurrent herpes simplex or (pre) cancerous lesions in the areas to be treated
* Known Diabetes mellitus or uncontrolled systemic diseases in the assessment of the investigator.
* Laser therapy, chemical peeling, dermabrasion or botulin toxin treatment in the area to be treated within less than three months prior to and during the course of the study.
* Current participation in another clinical investigation
* Subjects whose participation in clinical trials is prohibited by the Austrian Medical Devices Act (e.g, persons with a legal custodian appointed due to mental disability, prisoners, soldiers and other members of the armed forces, civil servants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Princess® RICH to correct fine lines on the face including lateral canthal lines (LCL) and perioral rhytids (PR) | Week 8 compared to Baseline
  Percentage of responders at week 8 Responder is defined as at least "improved" versus baseline in the fine lines of lateral canthal lines (LCL) and/or perioral rhytids (PR) assessed with the GAIS (Gloabel Aesthetic Improvement Scale)
  Global aesthetic improvement can be rated as 'very much improved', 'much improved', 'improved', 'no change' or 'worse

SECONDARY OUTCOMES:
Effectiveness of Princess® RICH to correct fine lines on the face including lateral canthal lines (LCL) and perioral rhytids (PR) | Week 12 and 16 compared to Baseline
  Percentage of responders at week 12 and 16.
Ability of Princess® RICH to improve skin hydration | Week 3, 6, 8, 12 and 16 compared to Baseline
  Change from baseline at weeks 3, 6, 8, 12 and 16 in skin hydration. Skin hydration is measured using a corneometer device.
Ability of Princess® RICH to improve skin tone | Week 3, 6, 8, 12 and 16 compared to Baseline
  Changes from baseline at weeks 3, 6, 8, 12 and 16 in skin tone. Skin tone is measured using a cutometer device.
Ability of Princess® RICH to improve skin elasticity | Week 3, 6, 8, 12 and 16 compared to Baseline
  Change from baseline at weeks 3, 6, 8, 12 and 16 in skin elasticity. Skin elasticity is measured using a cutometer device.
Subject satisfaction with treatment | Week 8, 12 and 16
  Subject satisfaction with treatment at weeks 8, 12 and 16. Satisfaction with the treatment will be graded using one of the following categories: "Very unsatisfied", "Unsatisfied", "Neither unsatisfied nor satisfied", "Satisfied", or "Very satisfied".

OTHER OUTCOMES:
Ocurrence and frequency of adverse events | Throughout the study (16 weeks)
  Assessment of occurrence and frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Monika Sulovsky, MD, Principal Investigator — Yuvell; Daisy Kopera, MD, Principal Investigator — Medizinische Universität Graz- Klinikum für Dermatologie und Venerologie; Thomas Rappl, MD, Principal Investigator — MaRa-Medical Aesthetic Research Academy
Locations (3):
- Austria (3):
  - MaRa-Medical Aesthetic Research Academy, Graz
  - Medizinische Universität-Klinikum für Dermatologie und Venerologie, Graz
  - YUVELL, Vienna